CLINICAL TRIAL: NCT05599074
Title: Treatment Results and Stability of Anterior Open Bite Cases Treated Using Extrusion Arches in Adults
Brief Title: Stability of Anterior Open Bite Treatment Using Extrusion Arches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Tasnim Yousry, Ms, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOBtreatmentinadults
Record Dates: First submitted 2022-10-18; First posted 2022-10-31 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Anterior Open Bite Malocclusion
Keywords: extrusion arches; anterior open bite; stability; extrusion; intrusion

STUDY DESIGN:
Intervention Model Description: Before and after design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AOB adults (Experimental): adult patients over 18 years having an anterior open bite of more than 2 mm, requiring incisors extrusion
  Interventions: Device: extrusion arch

INTERVENTIONS:
Device: extrusion arch — A stainless steel pre-formed arch wire custom made by placing V-bends 3-5 mm mesial to the molar tubes, placed into the auxiliary molar tubes after leveling phase and tied over the main arch wire distal to the lateral incisors

SUMMARY:
This study investigated treatment effects and stability of anterior open bite cases using extrusion arches

ELIGIBILITY:
Inclusion Criteria:

* adult patients above 18 years anterior open bite 2-6 mm full permanent dentition incisors requiring extrusion

Exclusion Criteria:

* increased incisal show at rest
* gum show at smiling cleft patients patient with tempro-mandibular joint problems FMA angle above 45

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
SNA angle | 18 months
  The anteroposterior position of maxillary base to the anterior cranial base.
SNB angle | 18 months
  The anteroposterior position of mandibular base to the anterior cranial base.
ANB angle | 18 months
  The anteroposterior position of maxillary base to the mandibular base.
SN-MP angle | 18 months
  Mandibular plane angle, the angle between the mandibular plane (Go-Me) and anterior cranial base plane (SN).
PP-MP angle | 18 months
  The angle between palatal plane (ANS-PNS) and mandibular plane.
AFH | 18 months
  Anterior facial height, the measurement between Nasion (N) and Menton (Me).
interincisal angle | 18 months
  - The inner angle between the long axis of the maxillary central incisor and long axis of mandibular central incisor.
L1 to MP in mm | 18 months
  - The perpendicular distance between the most anterior mandibular central incisor and mandibular plane.
L1 to MP angle | 18 months
  The angle between long axis of the most anterior central incisor and the mandibular plane.
overbite | 18 months
  Vertical distances between the incisal edges of the maxillary and mandibular central incisors, perpendicular to N-Me.
U1 to PP angular and linear measurements | 18 months
  -The angle and perpendicular distance between long axis of the most anterior upper central incisor and the Palatal plane (ANS-PNS).
u6 to pp angle | 18 months
  -The angle between the axis between mesial cusp tip and mesiobuccal root apex of the upper first molar and the palatal plane.
U6 to PP in mm | 18 months
  -The perpendicular distance between the mesial cusp tip of the upper first maxillary molar and the palatal plane.
L6 to MP angle | 18 months
  The angle between the axis between mesial cusp tip and mesial root apex of the lower first molar and the mandibular plane.
L6 to MP in mm | 18 months
  The perpendicular distance between mesial cusp tip of the lower first molar and the mandibular plane.

CONTACTS AND LOCATIONS:
Overall Officials: tasneem hammad, BDS, Principal Investigator — Alexandria University; hanan ismail, PHD, Study Director — Alexandria University
Locations (1):
- Alexandria faculty of Dentistry, Alexandria, Egypt